CLINICAL TRIAL: NCT01614353
Title: Medication-taking Preferences & Practices of Patients With Chronic Conditions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Washington State University (Other)
Collaborators: Providence Medical Research Center (Other)
Responsible Party: Principal Investigator, Roxanne Vandermause, Associate Professor, Washington State University
Other Study IDs: PI-12-001
Record Dates: First submitted 2012-06-01; First posted 2012-06-07 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Any Condition in N73.0 Specified as Chronic; Adult Disease; Pharmacological Action
Keywords: Multiple Chronic Conditions; Older Adults; New Prescription
MeSH Terms: conditions — Disease; Multiple Chronic Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Cohort: All participants (N=30) will be asked to identify perceptions and behaviors surrounding the medication-taking process using technology-assisted prompts and recordings. Half (n=15) of the participants will participate in two hermeneutic interviews using an interpretive phenomenological approach to generate an interpretation of the meaning of medication taking.
  Interventions: Other: Electronic Diaries; Other: Hermeneutic Interviews

INTERVENTIONS:
Other: Electronic Diaries — Participants (N=30) will maintain electronic diaries to record spontaneous thoughts and perceptions regarding the use of a newly prescribed drug over 30 days.
Other: Hermeneutic Interviews — Half of the enrolled participants (n=15) will participate in 2 hermeneutic interviews conducted in an interpretive phenomonological approach to generate an interpretation of the meaning of medication taking.

SUMMARY:
"Patients can easily be overwhelmed, confused and many times don't fully understand their need for new medications, or when the dosages are to be administered" (patient research partner quote). The long-term goal of this study is to refine medication science by developing patient-centered assessment, monitoring and management guidelines for patients and health professionals. The objective is to advance knowledge about the medication-taking perspectives, experiences, and behaviors of older adults with multiple chronic medical conditions (MCMC) to inform future research related to patient-centered medication prescribing, monitoring and management. This pilot study addresses the following PCORI interest area: "evaluating methods that can be used to assess the patient perspective when researching behaviors and choices within the patient's control that may influence outcomes." The rationale that underlies the proposed study is that medication-taking practices are wholly within patients' control, and are foundational to reducing complications and improving outcomes for those with MCMC. To meet the overall objective of this application, the following specific aims will be pursued: 1) identify perceptions and behaviors surrounding the medication-taking process of older adults with MCMC; and 2) generate an interpretation of the meaning of medication-taking among older adults with MCMC. To achieve these aims, data will be obtained in "real time" from patients (N=30) receiving a new prescription using smart phone technology. The smart phones will include prompts to help participants record thoughts about medication use throughout the day for 30 days. Findings from electronic diaries will be logged, analyzed and qualitatively analyzed. Some patients (n=15) will provide in-depth hermeneutic interviews to provide rich descriptions and interpretive commentary about the experience of receiving a new medication prescription. The objective is to uncover previously unidentified areas of common experience in older persons with multiple chronic conditions who have received a new prescription. Common experiences and patterns of influences, that are often surprising or unexpected, will be categorized and assessed. The expected outcomes of this pilot study are improved knowledge of medication-taking perceptions, experiences, and practices of older adults with MCMC-knowledge that is critical to advance patient-centered medication science.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Diagnosis of at least 3 chronic medical conditions
* Receiving 5 or more medications
* Receipt of a new prescription medication at enrollment
* Ability to speak English

Exclusion Criteria:

* Any individual that does not meet the 5 inclusion criteria listed above

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons seen at the Providence Kidney Disease and Hypertension Clinic, aged 60 years or older, with 3 chronic conditions, taking 5 or more medications, and who receive a prescription for a NEW medication will be invited to participate in the 30 day study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Identify perceptions and behaviors surrounding the medication-taking process of older adults with MCMC. | Daily electronic diaries for a duration of 30 days
  Data will be obtained in "real time" in that patients will audio record thoughts as they arise in the course of each day using an electronic device, over 30 consecutive days, and will answer questions related to medication use. Findings from end of day prompts will be logged using tables that compare participant demographic characteristics, whether or not the new medication or all prescribed medication was taken, and self-assessed level of wellness.
Generate an interpretation of the meaning of medication taking among older adults with MCMC. | 2 Interviews: 1 at enrollment and 1 at 30 days
  In-depth hermeneutic interviews and interpretive phenomenological analyses will be conducted for 15 of the 30 enrolled participants. Patterns and themes that capture common experiences revealed in these data provide language for further investigation and new discussion in areas that have been studied traditionally. Such findings are the characteristic "phenomenological contribution" of qualitative research. Interpretive commentary in the context of social and cultural evidence and extant literature on medication use will be generated.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Neumiller, PharmD, Principal Investigator — Washington State University; Roxanne Vandermause, PhD, Principal Investigator — Washington State University
Locations (2):
- United States (2):
  - Providence Medical Research Center, Spokane, Washington
  - Washington State University, Spokane, Washington